CLINICAL TRIAL: NCT02791815
Title: A Single-center, Open-label, Randomized, Two-treatment Crossover Study to Investigate the Effect of Selexipag on the Pharmacokinetics of Midazolam and Its Metabolite 1-hydroxymidazolam in Healthy Male Subjects
Brief Title: Potential Pharmacokinetic Interaction Between Selexipag and Midazolam in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AC-065-114; 2016-000856-83 (EudraCT Number)
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Subjects
Keywords: selexipag; pharmacokinetics; midazolam
MeSH Terms: interventions — Midazolam; selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): Subjects participate in two study periods: During the first period, they receive a single oral dose of midazolam on Day 1. During the second period, they receive oral selexipag alone from Day 1 to Day 11 and selexipag + midazolam on Day 12. There is a washout period of 14 to 21 days between the two periods.
  Interventions: Drug: Midazolam; Drug: Selexipag
- Sequence BA (Experimental): Subjects participate in two study periods: During the first period, they receive oral selexipag alone from Day 1 to Day 11 and selexipag + midazolam on Day 12. During the second period, they receive a single oral dose of midazolam on Day 1. There is a washout period of 14 to 21 days between the two periods.
  Interventions: Drug: Midazolam; Drug: Selexipag

INTERVENTIONS:
Drug: Midazolam — Single oral dose of 7.5 mg midazolam (tablet)
Drug: Selexipag — Oral administration of selexipag (200 µg film-coated tablet) for 12 consecutive days (with a titration scheme from 400 to 1600 μg b.i.d. )
  Other Names: ACT-293987

SUMMARY:
The primary purpose of this study is to evaluate the effect of repeated doses of selexipag on the pharmacokinetics of a single oral dose of midazolam (i.e., how long and how much midazolam is present in the blood)

DETAILED DESCRIPTION:
In order to exclude an inductive effect of selexipag in the gastrointestinal tract, this study aims at investigating the effect of selexipag on the PK of midazolam, a sensitive substrate of both hepatic and intestinal cytochrome P450 3A4 (CYP3A4).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent form
* Age from 18 to 45 years (inclusive) at screening
* Body mass index (BMI) from 18.0 to 28.0 kg/m2 (inclusive) at screening
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests

Key Exclusion Criteria:

* Any contraindication to the study treatments
* History or clinical evidence of any disease or medical / surgical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study treatments
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cmax of midazolam following administration of midazolam alone and in combination with selexipag | From pre-dose up to 24 hours after midazolam admisnitration for each treatment period
  Cmax is the maximum observed plasma concentration and is directly derived from the individual plasma concentration time curves of midazolam
AUC(0-inf) of midazolam following administration of midazolam alone and in combination with selexipag | From pre-dose up to 24 hours after midazolam admisnitration for each treatment period
  AUC(0-inf) is the area under the plasma concentration-time curves of midazolam, calculated from time 0 (pre-dose) to the extrapolated infinite time

SECONDARY OUTCOMES:
Cmax of 1-hydroxymidazolam following administration of midazolam alone and in combination with selexipag | From pre-dose up to 24 hours after midazolam admisnitration
AUC(0-inf) of 1-hydroxymidazolam following administration of midazolam alone and in combination with selexipag | From pre-dose up to 24 hours after midazolam admisnitration
tmax of midazolam and 1-hydroxymidazolam following administration of midazolam alone and in combination with selexipag | From pre-dose up to 24 hours after midazolam admisnitration
  tmax is the time to reach Cmax of midazolam and its metabolite (1-hydroxymidazolam), respectively
t½ of midazolam and 1-hydroxymidazolam following administration of midazolam alone and in combination with selexipag. | From pre-dose up to 24 hours after midazolam admisnitration
  t½ is the terminla half-life of midazolam and its metabolite (1-hydroxymidazolam), and corresponds to the period of time required for the concentration levels of midazolam and its metabolite to be reduced by one-half, respectively
Trough concentration of selexipag and its metabolite ACT-333679 at steady-state | Days 1, 4, 7, 10,12 and 13
  Trough concentrations are measured before morning administration of selexipag

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events and serious adverse events | Up to 39 days (from Day 1 of Period 1 to end of study of Period 2)
  A treatment-emergent AE is any AE temporally associated with the use of a study treatment, whether or not considered related to the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Eric Juif, PhD, Study Director — Actelion
Locations (1):
- Investigator Site, Gières, France